CLINICAL TRIAL: NCT03057457
Title: The NGAL Test™ As An Aid in the Risk Assessment for AKI Stage II and III in an Intensive Care Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioPorto Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: NGAL-001
Record Dates: First submitted 2017-02-13; First posted 2017-02-20 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Kidney Injury
  Interventions: Device: NGAL Test

INTERVENTIONS:
Device: NGAL Test — The purpose of this study is to demonstrate that BioPorto Diagnostic's NGAL test is able to assist in determining the risk for acute kidney injury for patients who have been admitted to the intensive care unit.

SUMMARY:
The NGAL TestTM is a particle-enhanced turbidimetric immunoassay for the quantitative determination of neutrophil gelatinase-associated lipocalin (NGAL) in human EDTA plasma for testing on automated clinical chemistry analyzer.

The First Indication for Use: An NGAL test result above the assay cutoff as an aid in the risk assessment for the development of stage II or III acute kidney injury (AKI) within 1 day of patient assessment in patients in the intensive care unit (ICU) who are hypotensive (MAP<70 mmHg) and/or receiving vasopressor support. Second Indication for Use: In patents with stage II or III AKI, NGAL measurement aids in the risk assessment of the development of persistent (≥2 days) stage 2 or 3 AKI.

The Primary Objective for this clinical trial is to validate that the NGAL test using a cutoff of 140 ng/ml shows clinical performance in predicting the development of moderate or severe acute kidney injury within 1 day. The Secondary Objective is to validate that the NGAL test shows clinical performance in predicting persistent moderate or severe acute kidney injury during any contiguous 2 day interval.

It is anticipated that up to 20 Clinical Sites in US will participate in the trial. The study sites will recruit consecutive patients meeting the inclusion and exclusion criteria who are admitted to hospital in an ICU or critical care setting. Patients will receive their clinical standard of care including standard laboratory and other testing as requested by each subject's physician.

DETAILED DESCRIPTION:
The NGAL TestTM is a particle-enhanced turbidimetric immunoassay for the quantitative determination of neutrophil gelatinase-associated lipocalin (NGAL) in human EDTA plasma for testing on automated clinical chemistry analyzer.

The First Indication for Use: An NGAL test result above the assay cutoff as an aid in the risk assessment for the development of stage II or III acute kidney injury (AKI) within 1 day of patient assessment in patients in the intensive care unit (ICU) who are hypotensive (MAP<70 mmHg) and/or receiving vasopressor support. Second Indication for Use: In patents with stage II or III AKI, NGAL measurement aids in the risk assessment of the development of persistent (≥2 days) stage 2 or 3 AKI.

The Primary Objective for this clinical trial is to validate that the NGAL test using a cutoff of 140 ng/ml shows clinical performance in predicting the development of moderate or severe acute kidney injury within 1 day. The Secondary Objective is to validate that the NGAL test shows clinical performance in predicting persistent moderate or severe acute kidney injury during any contiguous 2 day interval.

It is anticipated that up to 20 Clinical Sites in the US will participate in the trial. The study sites will recruit consecutive patients meeting the inclusion and exclusion criteria who are admitted to hospital in an ICU or critical care setting. Patients will receive their clinical standard of care including standard laboratory and other testing as requested by each subject's physician. Enrollment is estimated to take approximately six months and the trial will be stopped when the Adjudication Panel has diagnosed at least 85 patients with AKI stage 2 or 3.

Each subject who is enrolled in the study will only have 4 blood draws as part of NGAL TestTM Trial with no additional study activities with the exception of data collection. The NGAL results will not be returned to the treating physician for use in the health management of the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects should be enrolled within 24 hrs. of ICU admission, from ED or floor within 24 hrs. of ICU admission or if the subject is from another ICU no more than 24 hrs. from presentation.

  * Within 24 hrs. prior to enrollment the subject's

    o Cardiovascular SOFA score of >= 1(MAP<70 mmHg and/or receiving any vasopressor support
  * Subject or representative written informed consent
  * Subject > 18 years of age

Exclusion Criteria:

* If the subject is part of a special population (pregnancy, prisoners)
* If the subject has received a previous renal transplantation
* If the subject has been diagnosed with moderate to severe AKI prior to enrollment as defined by the treating physician (KDIGO Stage 2/3, RIFLE-I or RIFLE-F/AKIN 2 or AKIN 3) ,
* If the subject is currently on dialysis or in imminent need of dialysis at the time of enrollment
* The subject has been diagnosed with HIV or Hepatitis
* The subject has been diagnosed with Chronic Kidney disease without baseline value - CKD stage 4-5
* If the patient is on palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients diagnosed at high risk for developing AKI.
Sampling Method: Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | Up to 7 days in ICU or until discharge
  To demonstrate that the sum of sensitivity and specificity is greater than 1 using a cutoff of 140 ng/mL when compared to the primary clinical endpoint AKI as adjudicated KDIGO Stage 2/3 AKI

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado Kidney Care, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No